CLINICAL TRIAL: NCT04041011
Title: A Phase Ib Study of SHR-1316 in Combination With Fluzoparib（SHR-3162） in Small Cell Lung Cancer Patients
Brief Title: A Study of SHR-1316 and Fluzoparib（SHR-3162） in Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FZPL-Ib-106
Record Dates: First submitted 2019-07-31; First posted 2019-08-01 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1.Experimental: A (Part 1): Fluzoparib and SHR -1316 (Experimental)
  Interventions: Drug: 1.Experimental: A (Part 1): Fluzoparib and SHR -1316
- 2.Experimental: B (Part 1): Fluzoparib and SHR -1316 (Experimental)
  Interventions: Drug: 2.Experimental: B (Part 1): Fluzoparib and SHR -1316
- 3.Experimental: C (Part 2): Fluzoparib and SHR -1316 Expansion (Experimental)
  Interventions: Drug: 3.Experimental: C (Part 2): Fluzoparib and SHR -1316 Expansion

INTERVENTIONS:
Drug: 1.Experimental: A (Part 1): Fluzoparib and SHR -1316 — 1．Drug: Fluzoparib capsule will be given orally. Drug: SHR-1316 given intravenously (IV).
  Arms: 1.Experimental: A (Part 1): Fluzoparib and SHR -1316
Drug: 2.Experimental: B (Part 1): Fluzoparib and SHR -1316 — 2．Drug: Fluzoparib capsule will be given orally. Drug: SHR-1316 given intravenously (IV).
  Arms: 2.Experimental: B (Part 1): Fluzoparib and SHR -1316
Drug: 3.Experimental: C (Part 2): Fluzoparib and SHR -1316 Expansion — 3．Drug: Fluzoparib capsule will be given orally. Drug: SHR-1316 given intravenously (IV).
  Arms: 3.Experimental: C (Part 2): Fluzoparib and SHR -1316 Expansion

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of SHR-1316 in combination with Fluzoparib（SHR-3162） in Small Cell Lung Cancer Patients

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age.
* Histologically or cytologically confirmed SCLC.
* Failed at least one prior line of platinum-based chemotherapy.
* Patients must have measurable disease as defined by RECIST v1.1.
* ECOG 0-1.
* Adequate hematologic and organ function
* Signed inform consent form

Exclusion Criteria:

* Active or untreated central nervous system (CNS) metastases
* Spinal cord compression not definitively treated with surgery and/or radiation .
* Leptomeningeal disease
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Malignancies other than SCLC within 5 years prior to randomization
* History of autoimmune disease
* Positive test result for human immunodeficiency virus (HIV)
* Active hepatitis B or hepatitis C
* Severe infections
* Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of first administration of study treatment.
* Significant cardiovascular disease
* Prior allogeneic bone marrow transplantation or solid organ transplant
* Treatment with systemic immunosuppressive medications prior to randomization
* Pregnant or lactating women
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Part 1: 1.Number of Participants with AEs and SAEs | Up to approximately 24 months.
Part 1: 2. RP2D: Recommended dose for phase II study | Up to approximately 24 months.
Part 2: 1. ORR: Percentage of Participants With a CR or PR | Up to approximately 24 months.

SECONDARY OUTCOMES:
Part 1: 1. ORR: Percentage of Participants With a CR or PR | Up to approximately 24 months.
Part 2: 1.Number of Participants with AEs and SAEs | Up to approximately 24 months.
Part 2: 2.DoR: Percentage of Participants With a CR or PR | Up to approximately 24 months.
Part 2: 3. DCR: Percentage of participants in the analysis population who have a CR, PR or SD per RECIST 1.1. | Up to approximately 24 months.
Part 2: 4. PFS: PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first. | Up to approximately 24 months.
Part 2: 5. OS: Baseline until death from any cause | Up to approximately 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No